CLINICAL TRIAL: NCT02881671
Title: Identification of Genetic Basis of Atrioventricular Conduction Defects: From Congenital Forms to Degenerative Forms
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PROG/11/33
Record Dates: First submitted 2016-08-24; First posted 2016-08-29 (Estimated); Last update posted 2021-09-09 (Actual); Status verified 2021-09

CONDITIONS: Congenital Complete Heart Block; Cardiac Conduction Defect Progressive
Keywords: genetic; congenital atrioventricular block; progressive Cardiac Conduction Disease
MeSH Terms: conditions — Congenital heart block; Bundle-Branch Block

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Patients with congenital atrioventricular block: Patient with congenital atrioventricular block
  Interventions: Genetic: genetic blood analysis
- relatives with congenital atrioventricular block: Normal relatives of patients with congenital atrioventricular block
  Interventions: Genetic: genetic blood analysis
- Patients with progressive Cardiac Conduction Disease: Patients with progressive Cardiac Conduction Disease,
  Interventions: Genetic: genetic blood analysis
- relatives with progressive Cardiac Conduction disesae: Normal relatives of patients with progressive Cardiac Conduction Disease
  Interventions: Genetic: genetic blood analysis

INTERVENTIONS:
Genetic: genetic blood analysis — patients will undergo a blood sample (15 ml) to analyse their genetic profile

SUMMARY:
Identification of genes involved in congenital atrioventricular block and progressive Cardiac Conduction Disease.

DETAILED DESCRIPTION:
Atrioventricular blocks are a heterogenous group of diseases involving children with congenital atrioventricular block (CAB) and more frequently elderly patients affected by progressive Cardiac Conduction Disease (PCCD).

The aim of the study is to uncover the genetic model, likely more complex than previously appreciated, and characterize the gene expression remodelling leading to high degree of conduction defect.

The recent technological developments in genomics coupled to the availability of large and highly characterized biobanks of patients have now set the stage:

1. To identify rare genetic variants/new genes contributing to CAB and PCCD by exome sequencing on familial form suspected to impact strongly the phenotype
2. To identify common genetic variants modulating the risk of developing (severe) PCCD by GWAS
3. To estimate the prevalence and relevance of genes uncovered by TASK#1, #2 in large patient sets (PCCD and CAB) by NGS.

ELIGIBILITY:
Congenital atrioventricular block inclusion criteria:

* Patients with idiopathic congenital atrioventricular block diagnosed before the age of 15 years.
* Non-immune congenital atrioventricular block documented by a maternal serology (negative for anti-nuclear antibodies or anti Ro-SSA antibodies and anti La-SSB antibodies)
* Written consent to participate to the study and written consent of both parents.
* Parents of children with idiopathic congenital atrioventricular block.

Congenital atrioventricular block exclusion criteria

* Positive maternal serology
* Patients or parents who are unable to sign or who refuse to sign an informed consent

Progressive Cardiac Conduction Disease inclusion criteria

* Patients with isolated cardiac conduction disorder with a normal morphology of the heart confirmed by echocardiography.
* Relatives of patients with isolated cardiac conduction disorder
* Written consent to participate to the study

Progressive Cardiac Conduction Disease exclusion criteria

* Patients with cardiac conduction disorder associated with a structural cardiopathy or due to an identified cause
* Patients who are unable to sign or who refuse to sign an informed consent

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients of both sex with Atrioventricular Conduction Defects and relatives examined during familial screening
Sampling Method: Non-Probability Sample
Enrollment: 2600 (Estimated)
Dates: Start 2011-01 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Identification of genetic variations responsible of Atrioventricular Conduction Defects | inclusion

CONTACTS AND LOCATIONS:
Overall Officials: vincent PROBST, MD-PHD, Principal Investigator — Nantes University Hospital
Locations (2):
- France (2):
  - Chu Nantes, Nantes
  - Chu Rennes, Rennes

IPD SHARING:
Plan to Share IPD: No